CLINICAL TRIAL: NCT01410682
Title: Oral Care and Oropharyngeal and Tracheal Colonization by Gram-negative Pathogens in Children
Brief Title: Oral Care and Gram-negative Pathogen in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Mavilde da Luz Gonçalves Pedreira, Nursing School, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ORAL CARE
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-07

CONDITIONS: Tracheal and Oropharyngeal Colonization by Gram-negative Pathogens
Keywords: oral hygiene; ventilator-associated pneumonia; infection control; intensive care; pediatric nursing; pediatrics
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.12% Chlorhexidine Digluconate (Experimental): Oral care included use of an oral gel containing chlorhexidine digluconate 0.12% as an active ingredient (chlorhexidine digluconate 0.12%; methylcellulose gel 2.12%, 25 g; gooseberry syrup, 4 drops; menthol solution 50%,3 drops; and distilled water, to 30 g).The gel is applied on a toothbrush, and the teeth are cleaned in quadrants; all teeth surfaces are cleaned (vestibular,lingual, occlusal, and incisal). After each quadrant was cleaned, 10 mL of water (dispensed via a syringe) is used to rinse the quadrant and continual aspiration is used to remove all the gel and debris. After all the teeth are cleaned, the ventral surface of the tongue is brushed with posteriorto- anterior movements.
  Interventions: Other: 0,12% digluconate chlorhexidine
- tothbrushing (Placebo Comparator): This group received the same oral care that experimental group with the use of a similarly formulated gel without the antiseptic agent.The gel is applied on a toothbrush, and the teeth are cleaned in quadrants; all teeth surfaces are cleaned (vestibular, lingual, occlusal, and incisal). After each quadrant is cleaned, 10 mL of water (dispensed via a syringe) is used to rinse the quadrant and continual aspiration is used to remove all the gel and debris. After all the teeth are cleaned, the ventral surface of the tongue is brushed with posterior to anterior movements.
  Interventions: Other: toothbrushing

INTERVENTIONS:
Other: 0,12% digluconate chlorhexidine — Oral care with 0.12% Chlorhexidine Digluconate and toothbrushing is realized twice a day and took about 10 minutes to complete, depending on the child's acceptance and clinical conditions.
  Arms: 0.12% Chlorhexidine Digluconate
Other: toothbrushing — Gel is applied on a toothbrush, and the teeth are cleaned in quadrants; all teeth surfaces are cleaned (vestibular, lingual, occlusal, and incisal). After each quadrant is cleaned, 10 mL of water (dispensed via a syringe) is used to rinse the quadrant and continual aspiration is used to remove all the gel and debris. After all the teeth are cleaned, the ventral surface of the tongue is brushed with posterior to anterior movements.
  Arms: tothbrushing

SUMMARY:
Critical care nursing interventions related to oral care can reduce the microorganisms in the oropharynx available for translocation to other sites. THis is a randomized, controlled and double blinded study performed in a pediatric intensive care unit (PICU) from a Brazilian university hospital which objectives were to analyze 0.12% chlorhexidine digluconate influence on Gram-negative pathogens colonization of oropharyngeal and tracheal secretions of mechanically ventilated children.

ELIGIBILITY:
Inclusion Criteria:

* All the PICU children during 24 months of study were selected for participation.

Exclusion Criteria:

* newborns, those that fulfilled the Centers for Disease Control and Prevention criteria for pneumonia in infants and children at the time of PICU admission, PICU LOS less than 48 hours, presence of tracheostomy and those that declined to participate.

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Influence of chlorhexidine digluconate 0.12% on tracheal and oropharyngeal colonization by gram-negative pathogens

SECONDARY OUTCOMES:
Influence of some demographic characteristics of critically ill children on the oropharynx Gram-negative pathogens identification.